CLINICAL TRIAL: NCT05233787
Title: A Phase III Randomized Trial Evaluating the Tailored Versus the Systematic Use of Defunctioning Stoma After Total Mesorectal Excision for Rectal Cancer
Brief Title: Trial Evaluating the Tailored Versus the Systematic Use of Defunctioning Stoma After Total Mesorectal Excision for Rectal Cancer (GRECCAR17)
Acronym: GRECCAR17
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/10
Record Dates: First submitted 2021-11-08; First posted 2022-02-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer; Ileostomy; Functional Disturbance
Keywords: Rectal Cancer; Defunctioning stoma; Quality of life; Pelvic sepsis; Functional outcomes
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Tailored use of defunctioning stoma after TME (Experimental): The tailored use of defunctioning stoma includes two steps:
  * Firstly, the decision to use or not a defunctioning stoma will be based on the personalized risk of anastomotic leakage (according to AFOR score). This score is ranked from 0 to 6, and includes gender, Body Mass Index, smoking, diabetes, tumor size and preoperative radiotherapy.
  * Patients with AFORS equal to 0 or 1 (risk of anastomotic leakage less than 10%) will not have defunctioning stoma;
  * Patients with AFORS equal to or between 2 and 6 (risk of anastomotic leakage more than 20%) will have a defunctioning stoma.
  * Secondly, in patients with a defunctioning stoma, an early closure will be performed day 8-12 after TME if:
  * No fever postoperatively (≤ 38°C),
  * CRP at day 2 lower than 115mg/L (+/- 10 mg/L), decreasing at day 4,
  * CT-scan with colonic contrast retrograde enema showing no anastomotic leakage.
  Interventions: Procedure: Tailored use of defunctioning stoma after TME
- Arm B: Systematic use of defunctioning stoma (Active Comparator): Systematic use of defunctioning stoma for 3 months after TME according to French national guidelines
  Interventions: Procedure: Systematic use of defunctioning stoma

INTERVENTIONS:
Procedure: Tailored use of defunctioning stoma after TME — Tailored use of defunctioning stoma after TME based on a 2-step process:
  i) to perform or not a defunctioning stoma according to the personalized risk of anastomotic leakage (defunctioning stoma only if Anastomotic Failure Observed Risk Score=[2-6]), ii) to perform an early stoma closure at day 8-12, according to clinical (fever), biological (CRP level days 2 and 4 postoperatively) and radiological postoperative assessment (CT-scan with colonic contrast retrograde enema day 7-8 postoperatively)
  Arms: Arm A: Tailored use of defunctioning stoma after TME
Procedure: Systematic use of defunctioning stoma — Systematic use of defunctioning stoma for 2-3 months after TME, according to French national and international guidelines
  Arms: Arm B: Systematic use of defunctioning stoma

SUMMARY:
GRECCAR 17 will be the first prospective and randomized trial to assess a tailored policy in the use of defunctioning stoma after TME according to the personalized risk of anastomotic leakage. The tailored use of defunctioning stoma after TME for rectal cancer should improve both the quality of life of patients and the anorectal function, without any impact on anastomotic leakage. Moreover, for the healthcare system, this new approach could be a cost-effective strategy, leading to a decrease in healthcare expenses.

The main objective is to compare the impact of tailored defunctioning stoma after TME for rectal cancer versus the systematic use of defunctioning stoma on the evolution of the specific Quality Of Life (QLQC30) during the 12 months after surgery.

DETAILED DESCRIPTION:
The introduction of Total Mesorectal Excision (TME) as the surgical procedure of choice for low and mid rectal cancer has led to decrease local recurrence and improved oncological results. Postoperative morbidity remains a major issue, and the most feared complication is anastomotic leakage. The systematic use of a defunctioning stoma during 3 months to protect low colorectal anastomosis (below than 7 cm from the anal verge) is the standard of practice after TME surgery in order to decrease risks of anastomotic leakage and urgent re-operations.

However, there have been a lot of controversies surrounding the role of defunctioning stoma mainly due to stoma-related complications, ranked from 20% to 60%, which may lead to prolonged inpatient care, urgent re-operation and devastating effects on quality of life (QOL) and healthcare expenses. Moreover, it has been reported that patients either without defunctioning stoma, or with early stoma closure (days 8-12 after TME) have a better functional outcomes than patients with systematic defunctioning stoma for 3 months.

The experimental arm (arm A) will benefit from a tailored use of defunctioning stoma after TME based on a 2-step process: i) to perform or not a defunctioning stoma according to the personalized risk of anastomotic leakage (defunctioning stoma only if Anastomotic Failure Observed Risk Score=[2-6]), ii) to perform an early stoma closure at day 8-12, according to clinical (fever), biological (CRP level days 2 and 4 postoperatively) and radiological postoperative assessment (CT-scan with colonic contrast retrograde enema day 7-8 postoperatively). The control arm (arm B) will benefit from systematic use of defunctioning stoma for 2-3 months after TME, according to French national and international guidelines.

Patients will be followed at 1, 4, 8 and 12 months after surgery, with chest, abdominal and pelvic scan and tumour markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Rectal adenocarcinoma (histologically proven)
* No metastasis or medical history of colorectal metastasis (M0)
* Patients with rectal cancer < 12 cm from the anal verge (determined by rectal examination or MRI)
* Patients operated on by mini-invasive TME (laparoscopic, robotic or TaTME);
* With or without neo adjuvant treatment
* Realize a stapling anastomosis < 7 cm from the anal verge (determined by rectal examination or MRI)
* Patients with expected defunctioning ileostomy
* Appropriate hematologic function: hemoglobin ≥ 10.5 g/dL, leukocytes > 4000/mm3, blood platelets > 100,000/mm3);
* Appropriate renal function (serum creatinine < 15 mg/dL);
* Effective contraception of childbearing age : Male patients and premenopausal women should agree to use two medically validated contraceptive methods (one for the patient et one for the partner) during the study
* Patient affiliated or beneficiary to a health security system;
* Patient and doctor have signed informed consent

Exclusion Criteria:

* Patients with rectal cancer requiring TME surgery with handsewn anastomosis;
* Patients operated on by open approach;
* Previous pelvic irradiation for reasons other than rectal cancer
* Concomitant cancer or medical history of cancer within 5 years other than cancers treated in situ (cervical carcinoma or basocellular carcinoma or spinocellular carcinoma)
* Patients with expected defunctioning colostomy;
* Patients with perforated rectal cancer or preoperative pelvic sepsis;
* Patients with inflammatory bowel disease and/or bowel obstruction,
* Patients operated on in emergency;
* Patients with poor nutrition (Albumin < 34 g/L, pre-Alb < 0.14 g/L)
* Patients with extended-TME or pelvic exenteration (prostate);
* Patients with history of heart or vascular ischemia;
* Severe heart disease or congestive heart disease;
* Patients with immunodeficiency and/or under corticotherapy;
* Severe lung disease or respiratory failure;
* Severe kidney disease;
* Previous disease or disability expected to influence the assessment of postoperative QOL;
* Pregnancy or breast feeding;
* Persons deprived of liberty or under guardianship (curatorship or tutorship) or incapable of giving consent;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up scheduled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life over the 12 months after surgery | At 1, 4, 8, and 12 months of follow-up
  The QLQ-C30 is a patient self-rating questionnaire (30 questions) that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100 REF. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
  The area under the quality of life curve will be measured over the 12 months after rectal surgery, with measurement time points at 1, 4, 8 and 12 months.

SECONDARY OUTCOMES:
Proportion of anastomotic leakage | At 1 and 4 months after the rectal surgery
  Proportion of patients with an anastomotic leakage will be assessed by a clinical exam (with a rectal examination) at 1 month and with a clinical exam (with a rectal examination) and a CT scan at 4 months after rectal surgery
The PF, RF, CF, EF, SF, FA, PA, NV, QL Dimensions of the QLQ-C30 questionnaire | At 1, 4, 8 and 12 months after the rectal surgery
  1. 9 dimensions will be assessed with:
     * PF : Physical Functioning
     * RF : Role Functioning
     * CF : Cognitive Functioning
     * EF : Emotional Functioning
     * SF: Social Functioning
     * FA : Fatigue
     * PA : Pain
     * NV : Nausea and Vomiting
     * QL : Global health status
       2- The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. This is a patients self-rating questionnaire that measures five functional scales (physical, role, social, emotional, and cognitive) three symptom scales (fatigue, pain, nausea and vomiting) A global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. Scores can be linearly transformed to provide a score from 0 to 100 REF. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
The urinary frequency | At 1, 4, 8, and 12 months post-surgery
  The QLQ-CR29 (Quality of life of rectal cancer patients with 29 questions) has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items.
  Urinary frequency is measured with items 1 and 2 of the questionnaire. The score can range from 0 to 100.
  Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Blood or mucus in stools | At 1, 4, 8, and 12 months post-surgery
  The QLQ-CR29 (Quality of life of rectal cancer patients with 29 questions) has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items.
  The blood or mucus in stools is measured with items 8 and 9 of the questionnaire. The score can range from 0 to 50.
  Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Stool frequency | At 1, 4, 8, and 12 months post-surgery
Body image dimensions of the QLQ-CR29 questionnaire | At 1, 4, 8, and 12 months post-surgery
  The QLQ-CR29 (Quality of life of rectal cancer patients with 29 questions) has five functional and 18 symptom scales. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Rate of defunctioning stoma | At 1 month after the rectal surgery
  Proportion of patients who have a defunctioning stoma. It will be assessed at the time of the consultation at 1 month with the collection of the adverse events (AE) and the serious adverse events (SAE)
Low Anterior Resection Syndrome score (LARS score) | At 1, 4, 8 and 12 months after the rectal surgery
  The LARS questionnaire (low anterior resection score) evaluates bowel function. Five questions regarding incontinence for flatus and liquid stools, frequency, clustering and urgency for defecation are taken into account. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points).
Anal Incontinence (Wexner score) | At 1, 4, 8 and 12 months after the rectal surgery
  The WEXNER score assesses the importance of anal incontinence, it varies from 0 to 20, 20 corresponding to total anal incontinence
International Index of Erectile Function (IIEF)-5 | At 1, 4, 8 and 12 months after the rectal surgery
  Measured in male patients
Female Sexual Function Index (FSFI) scale scores | At 1, 4, 8 and 12 months after the rectal surgery
  Measured in female patients. The Female Sexual Function Index (FSFI) is a 19-item self-report inventory designed to assess female sexual function. It comprises six domains: desire, arousal ,lubrication orgasm, satisfaction, pain. The maximum score for each domain is 6.0, obtained by summing item responses and multiplying by a correction factor. The total composite sexual function score is a sum of domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0.
Urinary symptom profil (USP) | At 1, 4, 8, 12 months after the rectal surgery
  The Urinary symptom profil (USP) assesses urinary symptoms among men and women with stress, urge (from 0 to 9), overactive bladder (from 0 to 9), or urinary obstructive symptoms (from 0 to 9).
  The maximum corresponding to a bad result.
Postoperative morbidity (Clavien-Dindo score I-IV) | At 1 and 4 months after the rectal surgery
  This is a classification in order to rank a complication (surgical or medical morbidity) in an objective and reproducible manner.
  It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  It varies from 1 to 5, 5 corresponding to the death at the patient.
Postoperative mortality (Clavien-Dindo score V) | At 1 and 4 months after the rectal surgery
  This is a classification in order to rank a complication (surgical or medical morbidity) in an objective and reproducible manner.
  It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  It varies from 1 to 5, 5 corresponding to the death at the patient.
Proportion to work return after TME in active workers | Through study completion, an average of 1 year
  This endpoint is referring to the capability of active patients to resume their professional activity after surgery. In order to better describe this endpoint the investigators want to measure together the proportion of patients resuming their activity, and the time until resumption of professional activity.
Time to work return after TME in active workers | Through study completion, an average of 1 year
  This endpoint is referring to the capability of active patients to resume their professional activity after surgery. In order to better describe this endpoint the investigators want to measure together the proportion of patients resuming their activity, and the time until resumption of professional activity.
Quality of life over the 12 months after surgery | QLQ-C30 is assessed at 1, 4, 8 and 12 months after the rectal surgery
  The Quality of life of cancer contains 30 questions (QLQ-C30). This is a patients self-rating questionnaire that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100.Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Incremental cost-utility ratio defined as an incremental cost / Quality-Adjsuted Life Year (QALY) gained | From surgery to 12 months after surgery
  Costs will be measured through the French Health Data Hub database. QALYs will be measured using the and EQ-5D-5L questionnaire.
Total budgetary impact for French healthcare insurance system of spreading selective ostomy practice in France | From surgery to 12 months after surgery
  5-year financial model
Indirect Costs (€) for French Healthcare insurance scheme of sickness leaves | From surgery to 12 months after surgery
  Measured through SNDS database (Système National des Données de Santé) and data from our study on sickness leaves and times to return to work
Changes in microbiome composition and diversity from baseline to 1 month | From baseline to Month 1
  Data will be rarefied using the samples with the smallest number of reads and then subjected to alpha-diversity analysis employing Faith's phylogenetic diversity. Kruskal-Wallis will be calculated between all groups together and for pairwise comparisons. To find significant differences at the genera taxonomy level, ANCOM tests will be used to identify features that are differentially abundant across sample groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LAURENT, Principal Investigator — University Hospital, Bordeaux
Locations (28):
- France (28):
  - CHU Amiens-Picardie - Service de Chirurgie Digestive, Amiens
  - CHRU de Besançon - Service de Chirurgie Générale, Digestive et Cancérologique - Unité de Transplantation Hépatique, Besançon
  - CHU de Bordeaux - Service de Chirurgie Digestive et Endocrinienne - Unité Colorectale, Bordeaux
  - Clinique Tivoli Ducos - Service de Chirurgie Digestive, Bordeaux
  - CHU de Clermont-Ferrand - Service de Chirurgie Digestive et Hépato-biliaire, Clermont-Ferrand
  - APHP - Hôpital Beaujon - Service de Chirurgie Digestive, Clichy
  - CHU Grenoble Alpes - Service de Chirurgie Digestive, La Tronche
  - APHP - Hôpital Bicêtre - Service de Chirurgie Générale et Digestive, Le Kremlin-Bicêtre
  - CHU de Lille - Service de Chirurgie Générale et Digestive, Lille
  - Centre Lyonnais de Chirurgie Digestive, Lyon
  - APHM - Hôpital La Timone - Service de Chirurgie Digestive et Générale, Marseille
  - APHM - Hôpital Nord - Service de Chirurgie Digestive, Marseille
  - Hôpital Européen de Marseille - Service de Chirurgie Digestive, Marseille
  - Institut Paoli Calmette - Service de Chirurgie Digestive, Marseille
  - Institut du Cancer de Montpellier - Service de Chirurgie Digestive, Montpellier
  - APHP - HEGP- Service de Chirurgie Digestive, Paris
  - APHP - Hôpital Saint Antoine - Service de Chirurgie Digestive, Paris
  - APHP - Hôpital Saint-Louis - Service de Chirurgie Viscérale, Cancérologique et Endocrinienne, Paris
  - GH Diaconesses Croix Saint-Simon - Service de Chirurgie Digestive, Paris
  - Groupe Hospitalier Paris St. Joseph - Service de Chirurgie Digestive et Obésité, Paris
  - Hospices Civils de Lyon - Sevice de Chirurgie Digestive, Pierre-Bénite
  - CHU de Rennes - Service de Chirurgie Hépatobiliaire et Digestive, Rennes
  - CHU de Rouen - Service de Chirugie Digestive, Rouen
  - CHRU de Strasbourg - Service de Chirurgie Générale et, Strasbourg
  - CHU de Toulouse - Service de Chirurgie Digestive, Toulouse
  - CHRU de Tours - Service de Chirurgie Digestive Oncologique et Colorectale, Tours
  - CHRU de Nancy - Service de Chirugie Digestive, Hépatobiliaire, endocrinienne et Cancérologique, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy - Service de Chirurgie Viscérale Oncologique, Villejuif